CLINICAL TRIAL: NCT01040845
Title: A Pharmacokinetic Study to Evaluate the Effect of Colchicine on the Pharmacokinetic Profile of an Oral Contraceptive Containing Ethinyl Estradiol and Norethindrone in Healthy Women
Brief Title: A Pharmacokinetic Study of Colchicine With an Oral Contraceptive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MPC-004-07-1005
Record Dates: First submitted 2009-08-13; First posted 2009-12-30 (Estimated); Results first posted 2009-12-30 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-12

CONDITIONS: Pharmacokinetics
Keywords: healthy; pharmacokinetics; drug-interaction
MeSH Terms: interventions — ovcon 35; Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Contraceptive with Colchicine then Placebo (Experimental)
  Interventions: Drug: Norethindrone/Ethinyl Estradiol; Drug: Colchicine; Drug: Placebo (for Colchicine)
- Oral Contraceptive with Placebo then Colchicine (Placebo Comparator)
  Interventions: Drug: Norethindrone/Ethinyl Estradiol; Drug: Colchicine; Drug: Placebo (for Colchicine)

INTERVENTIONS:
Drug: Norethindrone/Ethinyl Estradiol — one tablet daily - 1 mg norethindrone/0.035 mg ethinyl estradiol on Days 1 to 21; inert ingredients on Days 22 to 28
Drug: Colchicine — 0.6mg tablet every 12 hours on Days 8 to 21
  Other Names: COLCRYS TM
Drug: Placebo (for Colchicine) — placebo tablet every 12 hours on Days 8 to 21

SUMMARY:
This study will evaluate the effect, if any, of twice daily dosing of colchicine 0.6 mg at steady state on the steady state pharmacokinetic profile of ethinyl estradiol and norethindrone (Ortho-Novum 1/35). It will also evaluate the effects, if any, of steady state ethinyl estradiol and norethindrone on colchicine at steady state. Finally, this study will assess the safety and tolerability of concurrent use of colchicine and an estrogen/progesterone-containing oral contraceptive.

DETAILED DESCRIPTION:
This study will evaluate the effect, if any, of twice daily dosing of colchicine 0.6 mg at steady state on the steady state pharmacokinetic profile of ethinyl estradiol and norethindrone (Ortho-Novum 1/35). It will also evaluate the effects, if any, of steady state ethinyl estradiol and norethindrone on colchicine at steady state. Finally, this study will assess the safety and tolerability of concurrent use of colchicine and an estrogen/progesterone-containing oral contraceptive. Following an optional single cycle run-in period in which subjects taking other oral contraceptives are switched to Ortho-Novum 1/35, 30 healthy adult female volunteers of child bearing age (18-45 years old) will be randomized in a double blind crossover fashion to receive each of two ethinyl estradiol and norethindrone dosing regimens in sequence. During each of the two dosing periods, subjects will receive one ethinyl estradiol and norethindrone tablet on the mornings of Days 1-7 of their cycles. On days 8-21, subjects will receive twice daily doses of either colchicine (0.6 mg capsule twice daily with breakfast and dinner) or the placebo (one capsule twice daily with breakfast and dinner), according to their randomization schedule, along with one ethinyl estradiol and norethindrone tablet. Subjects will receive the alternate dosing regimen in Cycle 2. Blood samples will be drawn at times sufficient to determine the steady state pharmacokinetics of ethinyl estradiol and norethindrone with and without steady state colchicine. In addition, during the cycle in which active colchicine is given, the effect of steady state ethinyl estradiol and norethindrone on steady state colchicine will be evaluated. Subjects will be monitored for adverse effects throughout the study via query and spontaneous reporting. Additionally baseline 12 lead EKG and vital signs will be compared to those obtained at time points throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking female volunteers of childbearing potential aged 18 to 45 years weighing at least 55 kg and within 15% of ideal body weight who are taking oral contraceptives on the advice of their personal health care provider and willing to switch to Ortho-Novum 1/35
* Subjects should be either sexually inactive or using a double barrier method of contraception for 14 days before the first dose of study drug and throughout the study

Exclusion Criteria:

* Pregnant or lactating
* Recent (2-year) history or evidence of alcoholism or drug abuse
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C antibody (HCV)
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease
* Hemoglobin < 12 g/dL
* Use of any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-gp within 30 days prior to the first dose of Ortho-Novum® 1/35 or expected to require such use

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty (30) healthy, non-smoking, premenopausal adult female volunteers, consisting of university students and members of the community at large, were to be enrolled.
Pre-assignment Details: 51 subjects screened, 21 were screen failures
Groups:
- Oral Contraceptive With Placebo Then Colchicine: [All subjects received each of the two study treatments in a randomly assigned sequence of two dosing cycles.] On the mornings of Days 1 to 20 of each cycle, each subject took one active tablet of Ortho-Novum 1/35. On Days 8 to 20, subjects additionally took one capsule of study drug (matching placebo capsule during the first cycle or over-encapsulated colchicine tablets 0.6 mg during the second cycle) twice daily. On Day 21 of each cycle, subjects received a single dose of study drug and a single active tablet of Ortho-Novum 1/35; then, 12 hours later, they received a second dose of study drug with a light snack. Inert Ortho-Novum 1/35 tablets were taken on Day 22 (after breakfast and the last blood sample), and then daily on Days 23 to 28.
- Oral Contraceptive With Colchicine Then Placebo: [All subjects received each of the two study treatments in a randomly assigned sequence of two dosing cycles.] On the mornings of Days 1 to 20 of each cycle, each subject took one active tablet of Ortho-Novum 1/35. On Days 8 to 20, subjects additionally took one capsule of study drug (over-encapsulated colchicine tablets 0.6 mg during or matching placebo capsule during the second cycle) twice daily. On Day 21 of each cycle, subjects received a single dose of study drug and a single active tablet of Ortho-Novum 1/35; then, 12 hours later, they received a second dose of study drug with a light snack. Inert Ortho-Novum 1/35 tablets were taken on Day 22 (after breakfast and the last blood sample), and then daily on Days 23 to 28.
Period: Overall Study
Arm/Group | Oral Contraceptive With Placebo Then Colchicine | Oral Contraceptive With Colchicine Then Placebo
Started | 15 | 15
Completed | 13 (withdrew consent due to schedule conflict (1); dropped by physician due to positive drug screen (1)) | 14 (withdrew consent due to schedule conflict (1))
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Oral Contraceptive With Placebo Then Colchicine; Oral Contraceptive With Colchicine Then Placebo: All subjects received each of the two study treatments in a randomly assigned sequence of two dosing cycles. On the mornings of Days 1 to 20 of each cycle, each subject took one active tablet of Ortho-Novum 1/35. On Days 8 to 20 of each cycle, subjects additionally took one capsule of study drug (either over-encapsulated colchicine tablets 0.6 mg or a matching placebo capsule) twice daily in the morning and with dinner. On Day 21 of each cycle, subjects received a single dose of study drug and a single active tablet of Ortho-Novum 1/35; then, 12 hours later, they received a second dose of study drug with a light snack. Inert Ortho-Novum 1/35 tablets were taken on Day 22 (after breakfast and the last blood sample).
- Total: Total of all reporting groups
Arm/Group | Oral Contraceptive With Placebo Then Colchicine | Oral Contraceptive With Colchicine Then Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants] — age range: >=18 and <=45
  Participants
    <=18 years | 0 | 0 | 0.0
    Between 18 and 65 years | 15 | 15 | 30.0
    >=65 years | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 23.8 (7.9) | 23.9 (4.2) | 23.9 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30.0
  Male | 0 | 0 | 0.0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0.0
  Asian | 0 | 0 | 0.0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0.0
  Black or African American | 0 | 0 | 0.0
  White | 15 | 15 | 30.0
  More than one race | 0 | 0 | 0.0
  Unknown or Not Reported | 0 | 0 | 0.0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30.0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration of Norethindrone With Colchicine at Steady State (Cmax, ss)
Description: The maximum or peak concentration that Norethindrone with Colchicine reaches in the plasma at steady state. Steady state refers to the point that constant concentration of drug is achieved subsequent to administration of constant doses of that drug given at constant intervals.
Time Frame: Day 21 of each cycle - plasma concentrations were drawn prior to the morning dose (0 hour) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 (prior to pm colchicine/placebo dose), and 24 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Norethindrone With Colchicine: On the mornings of Days 1 to 20, each subject took one active tablet of Ortho-Novum 1/35. On Days 8 to 20, subjects additionally took one colchicine tablet 0.6 mg (over-encapsulated to match placebo) twice daily, in the morning and with dinner. On Day 21, subjects received a single dose of colchicine 0.6 mg and a single active tablet of Ortho-Novum 1/35; then, 12 hours later, they received a second dose of colchicine 0.6 mg with a light snack. Inert Ortho-Novum 1/35 tablets were taken on Day 22 (after breakfast and the last blood sample), and then daily on Days 23 through 28.
Arm/Group | Norethindrone With Colchicine
Number analyzed (Participants) | 27
ng/mL | 24.17 (6.63)

2. Primary Outcome: Maximum Plasma Concentration of Norethindrone With Placebo at Steady State (Cmax, ss)
Description: The maximum or peak concentration that Norethindrone with Placebo reaches in the plasma at steady state. Steady state refers to the point that constant concentration of drug is achieved subsequent to administration of constant doses of that drug given at constant intervals.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Norethindrone With Placebo: On the mornings of Days 1 to 20, each subject took one active tablet of Ortho-Novum 1/35. On Days 8 to 20, subjects additionally took one placebo capsule twice daily in the morning and with dinner. On Day 21, subjects received a single dose of placebo and a single active tablet of Ortho-Novum 1/35; then, 12 hours later, they received a second dose of placebo with a light snack. Inert Ortho-Novum 1/35 tablets were taken on Day 22 (after breakfast and the last blood sample), and then daily on Days 23 through 28.
Arm/Group | Norethindrone With Placebo
Number analyzed (Participants) | 27
ng/mL | 24.42 (6.11)

3. Primary Outcome: Maximum Plasma Concentration of Ethinyl Estradiol With Colchicine at Steady State (Cmax, ss)
Description: The maximum or peak concentration that Ethinyl Estradiol with Colchicine reaches in the plasma at steady state. Steady state refers to the point that constant concentration of drug is achieved subsequent to administration of constant doses of that drug given at constant intervals.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ethinyl Estradiol With Colchicine: On the mornings of Days 1 to 20, each subject took one active tablet of Ortho-Novum 1/35. On Days 8 to 20, subjects additionally took one colchicine tablet 0.6 mg (over-encapsulated to match placebo) twice daily, in the morning and with dinner. On Day 21, subjects received a single dose of colchicine 0.6 mg and a single active tablet of Ortho-Novum 1/35; then, 12 hours later, they received a second dose of colchicine 0.6 mg with a light snack. Inert Ortho-Novum 1/35 tablets were taken on Day 22 (after breakfast and the last blood sample), and then daily on Days 23 through 28.
Arm/Group | Ethinyl Estradiol With Colchicine
Number analyzed (Participants) | 27
ng/mL | 0.14 (0.05)

4. Primary Outcome: Maximum Plasma Concentration of Ethinyl Estradiol With Placebo at Steady State (Cmax, ss)
Description: The maximum or peak concentration that Ethinyl Estradiol with Placebo reaches in the plasma at steady state. Steady state refers to the point that constant concentration of drug is achieved subsequent to administration of constant doses of that drug given at constant intervals.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ethinyl Estradiol With Placebo: On the mornings of Days 1 to 20, each subject took one active tablet of Ortho-Novum 1/35. On Days 8 to 20, subjects additionally took one placebo capsule twice daily in the morning and with dinner. On Day 21, subjects received a single dose of placebo and a single active tablet of Ortho-Novum 1/35; then, 12 hours later, they received a second dose of placebo with a light snack. Inert Ortho-Novum 1/35 tablets were taken on Day 22 (after breakfast and the last blood sample), and then daily on Days 23 through 28.
Arm/Group | Ethinyl Estradiol With Placebo
Number analyzed (Participants) | 27
ng/mL | 0.15 (0.05)

5. Primary Outcome: Maximum Plasma Concentration of Colchicine With Norethindrone/Ethinyl Estradiol at Steady State (Cmax, ss)
Description: The maximum or peak concentration that Colchicine with Norethindrone/Ethinyl Estradiol reaches in the plasma at steady state. Steady state refers to the point that constant concentration of drug is achieved subsequent to administration of constant doses of that drug given at constant intervals
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Colchicine With Norethindrone/Ethinyl Estradiol: On the mornings of Days 1 to 20, each subject took one active tablet of Ortho-Novum 1/35. On Days 8 to 20, subjects additionally took one colchicine tablet 0.6 mg (over-encapsulated to match placebo) twice daily, in the morning and with dinner. On Day 21, subjects received a single dose of colchicine 0.6 mg and a single active tablet of Ortho-Novum 1/35; then, 12 hours later, they received a second dose of colchicine 0.6 mg with a light snack. Inert Ortho-Novum 1/35 tablets were taken on Day 22 (after breakfast and the last blood sample), and then daily on Days 23 through 28.
Arm/Group | Colchicine With Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 27
ng/mL | 3.11 (0.86)

6. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)] for Norethindrone With Colchicine
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Norethindrone With Colchicine
Number analyzed (Participants) | 27
ng-hr/mL | 175.57 (60.74)

7. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)] for Norethindrone With Placebo
Description: as for outcome 6
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Norethindrone With Placebo
Number analyzed (Participants) | 27
ng/mL | 178.08 (51.69)

8. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)] Ethinyl Estradiol With Colchicine
Description: as for outcome 6
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.5, 5, 5.5, 6, 7, 8, 10, 14, 18, 24, 36, and 48 hours after drug administration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ethinyl Estradiol With Colchicine
Number analyzed (Participants) | 27
ng/mL | 1.24 (0.41)

9. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)] for Ethinyl Estradiol With Placebo
Description: as for outcome 6
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ethinyl Estradiol With Placebo
Number analyzed (Participants) | 27
ng/mL | 1.29 (0.40)

10. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)] for Colchicine With Norethindrone/Ethinyl Estradiol
Description: as for outcome 6
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Colchicine With Norethindrone/Ethinyl Estradiol
Number analyzed (Participants) | 27
ng/mL | 18.40 (4.15)

ADVERSE EVENTS:
Groups:
- Oral Contraceptive With Colchicine: On the mornings of Days 1 to 20, each subject took one active tablet of Ortho-Novum 1/35. On Days 8 to 20 of each cycle, subjects additionally took one colchicine tablet 0.6 mg (over-encapsulated to match placebo) twice daily, in the morning and with dinner. On Day 21 of each cycle, subjects received a single dose of colchicine 0.6 mg and a single active tablet of Ortho-Novum 1/35; then, 12 hours later, they received a second dose of colchicine 0.6 mg with a light snack. Inert Ortho-Novum 1/35 tablets were taken on Day 22 (after breakfast and the last blood sample), and then daily on Days 23 through 28.
Arm/Group | Oral Contraceptive With Colchicine
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 10
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Oral Contraceptive With Colchicine
eye pain (Eye disorders) | 1/27 (1)
eye discharge (Eye disorders) | 1/27 (1)
ocular hyperaemia (Eye disorders) | 1/27 (1)
abdominal pain upper (Gastrointestinal disorders) | 3/27 (3)
diarrhoea (Gastrointestinal disorders) | 5/27 (5)
nausea (Gastrointestinal disorders) | 3/27 (3)
stomach discomfort (Gastrointestinal disorders) | 1/27 (1)
fatigue (General disorders) | 1/27 (1)
feeling hot (General disorders) | 1/27 (1)
paronychia (Infections and infestations) | 1/27 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1/27 (1)
dizziness (Nervous system disorders) | 1/27 (1)
syncope (Nervous system disorders) | 1/27 (1)
metrorrhagia (Reproductive system and breast disorders) | 1/27 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/27 (1)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/27 (1)
cold sweat (Skin and subcutaneous tissue disorders) | 2/27 (2)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/27 (1)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1/27 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days